CLINICAL TRIAL: NCT05097534
Title: A Comprehensive Community Approach for Diabetes Prevention and Care for a Vulnerable Population in Galveston
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-0194
Record Dates: First submitted 2021-09-22; First posted 2021-10-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iDSMES (Active Comparator): Eligible study subjects randomized to the intervention arm will receive:
  A. Intensive Diabetes Self-Management, Education, and Support (iDSMES). Participants will be enrolled in groups in a virtual or in-person setting with their lifestyle coach, in this one-year educational program B. Services addressing Social Determinants of Health All study subjects will have their data collected at time points around baseline, 6 months and 12 months from consenting including glycemic control, hypertension management, dyslipidemia management, prevention or management of complications, healthcare outcomes, lifestyle change outcomes, patient-centeredness outcomes, Secondary diabetes self-management behaviors, self-efficacy in managing diabetes, diabetes distress, and Morisky Green Levine Medication Adherence Scale.
  Interventions: Other: iDSMES
- Standard of Care (Placebo Comparator): Eligible study subjects randomized to the intervention arm will receive standard of care offered to patients with diabetes.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: iDSMES — Intensive Diabetes Self-Management Education and Support combined with Addressing Social Determinants of Health
  Arms: iDSMES
Other: Standard of Care — Standard of Care for patients with type 2 diabetes
  Arms: Standard of Care

SUMMARY:
To improve diabetes self-management outcomes, patients with type 2 diabetes (n=150 - aged 13-84) recruited from St. Vincent Clinic (SVC) and Teen Health Center Inc., Clinics will be randomized using block randomization to receive standard of care or the integrated model. Patients in the intervention arm will be assessed for social and physical needs before being enrolled in a year-long education program (iDSMES). Enrollees will receive dietary counseling, physical and occupational therapy, in addition to other mental, financial and social benefits counseling. The investigators will compare the intervention outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 13-84, and
2. Patients diagnosed with type 2 diabetes, and
3. Patients have a BMI equal to or >25 (23, if Asians), and
4. Hemoglobin A1c value equal to or >7%

Exclusion Criteria:

1. Ages <13 or >84
2. Pregnancy. If a subject becomes pregnant, they will advised to discontinue the study.
3. Previous diagnosis of type 1 diabetes
4. Inability to participate for 12-month duration (e.g., Disorders that might compromise survival, planning to relocate outside the geographical coverage of University of Texas Medical Branch (UTMB) clinics
5. Other medical condition or medication administration deemed exclusionary by the study investigators
6. Prisoners

Ages: 13 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline HbA1c | at 6 months
  measurement of hemoglobin A1c (HbA1c %)
Change from baseline HbA1c | at 12 months
  measurement of hemoglobin A1c (HbA1c %)

SECONDARY OUTCOMES:
Change from baseline weight | at 6 months
  measurement of body weight in Kg
Change from baseline weight | at 12 months
  measurement of body weight in Kg
Change from baseline blood pressure | at 6 months
  measurement of systolic and diastolic blood pressure in mm Hg
Change from baseline blood pressure | at 12 months
  measurement of systolic and diastolic blood pressure in mm Hg
Change from baseline lipid profile | at 6 months
  measurement of lipid profile: Total Cholesterol, Triglycerides, High-Density Lipoprotein, and Low-Density Lipoprotein in mg/dL
Change from baseline lipid profile | at 12 months
  measurement of lipid profile: Total Cholesterol, Triglycerides, High-Density Lipoprotein, and Low-Density Lipoprotein in mg/dL
Change from baseline frequency of provider encounter | at 6 months
  Frequency of provider encounter
Change from baseline frequency of provider encounter | at 12 months
  Frequency of provider encounter
Change from baseline frequency of feet examination for neuropathy | at 6 months
  Frequency of feet examination for neuropathy
Change from baseline frequency of feet examination for neuropathy | at 12 months
  Frequency of feet examination for neuropathy
Change from baseline frequency of urine exam for microalbuminuria | at 6 months
  Frequency of urine exam for microalbuminuria
Change from baseline frequency of urine exam for microalbuminuria | at 12 months
  Frequency of urine exam for microalbuminuria
Change from baseline frequency of oral health checkup | at 6 months
  Frequency of oral health checkup
Change from baseline frequency of oral health checkup | at 12 months
  Frequency of oral health checkup
Change from baseline frequency of eye fundus examination | at 6 months
  Frequency of eye fundus examination
Change from baseline frequency of eye fundus examination | at 12 months
  Frequency of eye fundus examination
Change from baseline frequency of emergency care visits for treatment of T2-related issues | at 6 months
  Frequency of emergency care visits for treatment of T2-related issues
Change from baseline frequency of emergency care visits for treatment of T2-related issues | at 12 months
  Frequency of emergency care visits for treatment of T2-related issues
Change from baseline frequency of hospitalizations and re-admissions | at 6 months
  Frequency of hospitalizations and re-admissions
Change from baseline frequency of hospitalizations and re-admissions | at 12 months
  Frequency of hospitalizations and re-admissions
Participation in iDSMES classes (for those in the intervention arm only) | at 12 months
  Participation in iDSMES classes (total number of sessions attended)
Lifestyle change outcomes (for those in the intervention arm only) | every session through study completion, an average of 1 year
  Physical activity minutes in the last week prior to session
Change from baseline patient-centeredness | at 6 months
  General self-rated Health (GSRH): a single item survey- self-administered single question such as "in general, would you say that your health is? excellent, very good, good, fair, or poor?", where excellent is scored as "5" and poor is scored as "0".
Change from baseline patient-centeredness | at 12 months
  General self-rated Health (GSRH): a single item survey- self-administered single question such as "in general, would you say that your health is? excellent, very good, good, fair, or poor?", where excellent is scored as "5" and poor is scored as "0".
Change from baseline secondary diabetes self-management behaviors | at 6 months
  fifty-six-item survey. This includes a series of secondary diabetes self-management behaviors to explore mediating factors that might influence changes in glycemic control. We will assess the proportion of individuals with severe hypoglycemic episodes and use the brief modified Block seven-item diet screener with a four-week time horizon to determine the number of servings per day of fruit and vegetables.
Change from baseline secondary diabetes self-management behaviors | at 12 months
  fifty-six-item survey. This includes a series of secondary diabetes self-management behaviors to explore mediating factors that might influence changes in glycemic control. We will assess the proportion of individuals with severe hypoglycemic episodes and use the brief modified Block seven-item diet screener with a four-week time horizon to determine the number of servings per day of fruit and vegetables.
Change from baseline self-efficacy in managing diabetes | at 6 months
  This self-management resource center validated eight-item survey on patient confidence in performing certain activities. The survey is scored from 0 to 10 on a visual analog scale (VAS).
Change from baseline self-efficacy in managing diabetes | at 12 months
  This self-management resource center validated eight-item survey on patient confidence in performing certain activities. The survey is scored from 0 to 10 on a visual analog scale (VAS).
Change from baseline diabetes distress | at 6 months
  a two-item screening tool on 17 potential problems in the life of patients with diabetes. Patients are asked to score the distress ensuing from each problem during the last month from 1 to 6, where 1 is "Not a problem" and 6 is "a very serious problem".
Change from baseline diabetes distress | at 12 months
  a two-item screening tool on 17 potential problems in the life of patients with diabetes. Patients are asked to score the distress ensuing from each problem during the last month from 1 to 6, where 1 is "Not a problem" and 6 is "a very serious problem".
Change from baseline medication Adherence | at 6 months
  "Morisky Green Levine" Medication Adherence Scale: a four-item tool queries about forgetfulness, carelessness, and feelings around taking medications, scored from 0 to 4.
Change from baseline medication Adherence | at 12 months
  "Morisky Green Levine" Medication Adherence Scale: a four-item tool queries about forgetfulness, carelessness, and feelings around taking medications, scored from 0 to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent House Clinic, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes